CLINICAL TRIAL: NCT01675661
Title: Achieving Cannabis Cessation: Evaluating N-Acetylcysteine Treatment (ACCENT)
Brief Title: Achieving Cannabis Cessation-Evaluating N-Acetylcysteine Treatment
Acronym: ACCENT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kevin Gray, MD, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTN-0053; U10DA013727 (NIH); UG1DA013727 (NIH); U10DA013045 (NIH); U10DA015815 (NIH); U10DA013732 (NIH); U10DA015831 (NIH); U10DA020024 (NIH)
Record Dates: First submitted 2012-08-19; First posted 2012-08-30 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-04

CONDITIONS: Cannabis Dependence
MeSH Terms: conditions — Marijuana Abuse | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NAC plus CM (Active Comparator): N-acetylcysteine (NAC) plus Contingency Management (CM)
  Interventions: Drug: N-Acetylcysteine
- Placebo plus CM (Placebo Comparator): Placebo plus Contingency Management (CM)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-Acetylcysteine — Study participants randomly assigned to the NAC arm will receive a 12-week course of N-Acetylcysteine (1200mg) twice daily. All participants will concurrently participate in weekly medication management sessions and twice-weekly contingency management interventions.
  Other Names: NAC
  Arms: NAC plus CM
Drug: Placebo — Study participants randomly assigned to the placebo arm will receive a matched placebo twice daily. All participants will concurrently participate in weekly medication management sessions and twice-weekly contingency management interventions.
  Arms: Placebo plus CM

SUMMARY:
The primary objective of this study is to evaluate the impact of N-acetylcysteine (NAC) 1200 mg versus matched placebo (PBO) twice daily, added to contingency management (CM), on cannabis use among treatment-seeking cannabis-dependent adults (ages 18-50).

DETAILED DESCRIPTION:
The primary objective of this Phase 3 study is to evaluate the impact of NAC 1200 mg versus matched placebo (PBO) twice daily, added to contingency management (CM), on cannabis use among treatment-seeking cannabis-dependent adults (ages 18-50). After assessment and inclusion into the study, participants will be randomized to receive a 12-week course of NAC 1200 mg or matched placebo twice daily. All participants will concurrently participate in a twice-weekly contingency management (CM) intervention. Medication management will be conducted weekly throughout treatment by the medical clinician. Urine cannabinoid testing will occur at all visits, and will be used as the primary determinant of cannabis use. Participants will return approximately four weeks after treatment conclusion for evaluation of adverse events with medication discontinuation and sustained treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Must be able to understand the study and provide written informed consent
* Must meet current DSM-IV criteria for cannabis dependence in the last 30 days
* Must express interest in treatment for cannabis dependence
* Must submit a positive urine cannabinoid test during screening
* Women of child bearing potential must agree to use appropriate birth control methods during study participation: oral contraceptives, contraceptive patch, barrier (diaphragm or condom), levonorgestrel implant, medroxyprogesterone acetate, complete abstinence from sexual intercourse, or hormonal contraceptive vaginal ring

Exclusion Criteria:

* Allergy or intolerance to N-Acetylcysteine
* Women who are pregnant or lactating
* Current use of NAC or any supplement containing N-Acetylcysteine (must agree not to take any such supplement throughout study participation)
* Use of carbamazepine or nitroglycerin within 14 days of randomization
* Current enrollment in treatment for cannabis dependence
* Any use of synthetic cannabinoids (such as K2/Spice) in the 30 days prior to screening or during the period between screening and randomization
* Current substance dependence, other than cannabis or nicotine
* Urine drug screen positive for any drug of abuse other than cannabis or amphetamines at the randomization visit (Only participants who have a valid prescription for amphetamines (e.g., for ADHD) may be included)
* Urine drug screen positive for amphetamines at the randomization visit without having a valid prescription for it
* Maintenance treatment with buprenorphine or methadone
* Recent history of asthma (within the last 3 years)
* History of seizure disorder, bipolar disorder, schizophrenia, or other significant or unstable medical or psychiatric illness that may place the participant at increased risk in the judgment of the medical clinician
* Significant risk of homicide or suicide

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 302 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Gray, MD, Principal Investigator — Associate Professor, Department of Psychiatry and Behavioral Sciences, Medical University of South Carolina
Locations (6):
- United States (6):
  - UCLA Integrated Substance Abuse Programs, Los Angeles, California
  - APT Foundation, Inc., New Haven, Connecticut
  - University of Kentucky, Lexington, Kentucky
  - CODA, Inc., Portland, Oregon
  - Behavioral Health Services of Pickens County, Pickens, South Carolina
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
The lead investigator will submit coded individual level data on Clinical Trials Network (CTN) study participants to the Data Management Center contracted by NIDA Center for CTN. These data may include but are not limited to: demographic information, date of birth, medical history, substance use history, psychiatric history, objective measures of substance use and psychiatric status, HIV status and genetic information. Data will be submitted without information that could readily identify the study participant (i.e. We will not share medical record numbers, social security numbers or participant names or phone numbers with the Data Management Center). De-identified data will be made publicly available per the CTN's policies.

REFERENCES:
- [Background] McClure EA, Sonne SC, Winhusen T, Carroll KM, Ghitza UE, McRae-Clark AL, Matthews AG, Sharma G, Van Veldhuisen P, Vandrey RG, Levin FR, Weiss RD, Lindblad R, Allen C, Mooney LJ, Haynes L, Brigham GS, Sparenborg S, Hasson AL, Gray KM. Achieving cannabis cessation -- evaluating N-acetylcysteine treatment (ACCENT): design and implementation of a multi-site, randomized controlled study in the National Institute on Drug Abuse Clinical Trials Network. Contemp Clin Trials. 2014 Nov;39(2):211-23. doi: 10.1016/j.cct.2014.08.011. Epub 2014 Aug 30. PMID 25179587
- [Derived] Borodovsky JT, Sofis MJ, Sherman BJ, Gray KM, Budney AJ. Characterizing cannabis use reduction and change in functioning during treatment: Initial steps on the path to new clinical endpoints. Psychol Addict Behav. 2022 Aug;36(5):515-525. doi: 10.1037/adb0000817. Epub 2022 Jan 27. PMID 35084903
- [Derived] Sherman BJ, Sofis MJ, Borodovsky JT, Gray KM, McRae-Clark AL, Budney AJ. Evaluating cannabis use risk reduction as an alternative clinical outcome for cannabis use disorder. Psychol Addict Behav. 2022 Aug;36(5):505-514. doi: 10.1037/adb0000760. Epub 2021 Jul 1. PMID 34197135
- [Derived] Tomko RL, Baker NL, Hood CO, Gilmore AK, McClure EA, Squeglia LM, McRae-Clark AL, Sonne SC, Gray KM. Depressive symptoms and cannabis use in a placebo-controlled trial of N-Acetylcysteine for adult cannabis use disorder. Psychopharmacology (Berl). 2020 Feb;237(2):479-490. doi: 10.1007/s00213-019-05384-z. Epub 2019 Nov 11. PMID 31712969
- [Derived] Hser YI, Mooney LJ, Huang D, Zhu Y, Tomko RL, McClure E, Chou CP, Gray KM. Reductions in cannabis use are associated with improvements in anxiety, depression, and sleep quality, but not quality of life. J Subst Abuse Treat. 2017 Oct;81:53-58. doi: 10.1016/j.jsat.2017.07.012. Epub 2017 Jul 29. PMID 28847455
- [Derived] Gray KM, Sonne SC, McClure EA, Ghitza UE, Matthews AG, McRae-Clark AL, Carroll KM, Potter JS, Wiest K, Mooney LJ, Hasson A, Walsh SL, Lofwall MR, Babalonis S, Lindblad RW, Sparenborg S, Wahle A, King JS, Baker NL, Tomko RL, Haynes LF, Vandrey RG, Levin FR. A randomized placebo-controlled trial of N-acetylcysteine for cannabis use disorder in adults. Drug Alcohol Depend. 2017 Aug 1;177:249-257. doi: 10.1016/j.drugalcdep.2017.04.020. Epub 2017 Jun 10. PMID 28623823

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred almost exclusively through advertising. Individuals currently in treatment for cannabis dependence were not eligible to participate
Period: Overall Study
Arm/Group | NAC Plus CM | Placebo Plus CM
Started | 153 | 149
Completed | 113 | 103
Not Completed | 40 | 46
Not completed — Lost to Follow-up | 22 | 23
Not completed — Practical problems | 9 | 5
Not completed — Moved away | 5 | 6
Not completed — Withdrawal by Subject | 3 | 7
Not completed — Physician Decision | 0 | 2
Not completed — Death | 0 | 1
Not completed — Other reason | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NAC Plus CM | Placebo Plus CM | Total
Number analyzed (Participants) | 153 | 149 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (8.74) | 30.8 (9.32) | 30.3 (9.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 50 | 86
  Male | 117 | 99 | 216
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 34 | 65
  Not Hispanic or Latino | 122 | 115 | 237
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 44 | 40 | 84
  White | 84 | 92 | 176
  More than one race | 13 | 6 | 19
  Unknown or Not Reported | 10 | 7 | 17
Region of Enrollment [Number; unit: participants]
  United States | 153 | 149 | 302

OUTCOME MEASURES:

1. Primary Outcome: The Odds of Negative Urine Cannabinoid Tests During Treatment.
Description: The primary outcome is the abstinence rate over the 12 weeks of treatment. Abstinence is based on a weekly urine drug screen confirmed by central laboratory testing and defined as a negative cannabinoid result.
Time Frame: study weeks 2-13
Population: Intent to treat; all participants randomized
Measure: Number; unit: cannabis negative urine tests
Arm/Group | NAC Plus CM | Placebo Plus CM
Number analyzed (Participants) | 153 | 149
cannabis negative urine tests
  Study Week 2 | 25 | 21
  Study Week 3 | 30 | 22
  Study Week 4 | 33 | 36
  Study Week 5 | 32 | 33
  Study Week 6 | 32 | 30
  Study Week 7 | 36 | 37
  Study Week 8 | 40 | 37
  Study Week 9 | 39 | 36
  Study Week 10 | 39 | 37
  Study Week 11 | 38 | 36
  Study Week 12 | 34 | 40
  Study Week 13 | 33 | 36
  Overall | 410 | 401
Statistical Analysis 1: Comparison: NAC Plus CM vs Placebo Plus CM; For the primary outcome measure, a repeated-measures logistic regression model was used to analyze the odds of a negative urine cannabinoid test as an indicator of abstinence across all 12 weeks of treatment. A generalized estimating equations (GEEs) were used to adjust for this correlation with multiple samples per participant. The model for the primary analysis included the main effect of treatment, main effect of time, site effects, effect of smoking tobacco, and timeXtreatment interaction; Test type: Superiority or Other; p = 0.985, Regression, Logistic; OR=1.00; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.63 to 1.59]

ADVERSE EVENTS:
Time Frame: Evaluation of adverse events began after informed consent and continued at each weekly visit until the final 13 week follow up visit for all participants.
Description: Participants were asked once a week
Arm/Group | NAC Plus CM | Placebo Plus CM
Serious Adverse Events (participants affected / at risk) | 1/153 | 6/149
Other Adverse Events (participants affected / at risk) | 40/153 | 45/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAC Plus CM (N=153) | Placebo Plus CM (N=149)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Inpatient hospitalization for acute exacerbation of asthma
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) — Inpatient admission for lower extremity cellulitis-resolved without sequelae
Irregular Heart Rate (Cardiac disorders) | 0 (0) | 1 (1) — Inpatient admission for irregular heart beat; resolved without sequelae
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Inpatient hospitalization for herniated disc; resolved without sequelae
Dysfunctional Uterine Bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Inpatient hospitalization for dysfunctional uterine bleeding; resolved without sequelae
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Death due to motor vehicle accident
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) — Inpatient hospitalization for suicidal ideation; resolved without sequelae
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAC Plus CM (N=153) | Placebo Plus CM (N=149)
Nausea (Gastrointestinal disorders) | 7 (7) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 8 (8) | 8 (8)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Frequent Bowel Movements (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 10 (10) | 15 (15)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Elevated mood (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Human bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2)
Feeling abnormal (General disorders) | 0 (0) | 1 (1)
Energy increased (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Localized infection (Infections and infestations) | 0 (0) | 1 (1)
Groin Abscess (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications/dissemination products must be reviewed and approved by the Center for Clinical Trials Network (CCTN) Publications Committee before publishing/disseminating.